CLINICAL TRIAL: NCT06147726
Title: Effectiveness of Virtual Reality Supported Upper Extremity Position Matching Exercises in Parkinson's Disease Patients
Brief Title: Upper Extremity Rehabilitation With Virtual Reality in Parkinson's Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramazan KURUL (Other)
Collaborators: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor-Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Organization: Abant Izzet Baysal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-BENLI-005
Record Dates: First submitted 2023-09-27; First posted 2023-11-28 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease; Virtual Reality; Neurological Rehabilitation; Upper Extremity Dysfunction
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 2 groups, conventional physiotherapy to the control group
Who Masked: Outcomes Assessor
Masking Description: the physiotherapist administering the treatment and the physiotherapist performing the assessments will be different people
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Active Comparator): group to receive virtual reality supported upper extremity rehabilitation in addition to conventional physiotherapy
  Interventions: Other: Upper extremity position matching exercises in virtual reality; Other: Conventional physiotherapy
- Control group (Active Comparator): The group that will receive conventional physiotherapy for the total treatment time of the VR group
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Upper extremity position matching exercises in virtual reality — In addition to conventional treatment approaches for 20 minutes 2 days a week for 8 weeks, joint positioning exercises (4 different game sequences of 4 minutes, 1 minute rest between each sequence, total 20 minutes) designed specifically for the individual's existing range of motion will be applied to the VR group.
  Arms: VR group
Other: Conventional physiotherapy — proprioceptive neuromuscular facilitation techniques, parkinson-specific upper extremity and balance and gait exercises

SUMMARY:
Upper extremities are the first part of the body to be affected by Parkinson's disease. Although studies have shown that virtual reality-assisted rehabilitation methods are effective on gait and balance, studies on their use for upper extremity rehabilitation are limited. For this reason, the aim of the project is to examine whether virtual reality supported upper extremity position matching exercises, which will be specially prepared according to joint ranges of motion, will provide functional improvement in the upper extremities of individuals with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by motor disorders. Difficulties in using the upper limbs caused by these motor impairments are common with the disease. Upper limb motor impairments in PD include slowness of movement, difficulties in performing sequential tasks and limitations in upper limb function. Studies show that the upper extremities are usually the most affected body region in the early stages of PD. Despite this, the number of rehabilitation methods that can be used for upper extremity rehabilitation is limited. Impairments in upper extremity motor function constitute a leading problem in the lives of individuals with PD by affecting their ability to perform activities of daily living. Virtual reality applications stand out as an innovative approach in neurorehabilitation. Previous studies have reported positive effects of virtual reality on gait function and balance in PD. However, the number of studies designed with virtual reality for the upper limb is limited. Therefore, this project aims to fill the gap in the literature by examining the effectiveness of virtual reality-based rehabilitation in PD with a particular focus on upper extremity motor function and proprioception.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the research
* Being diagnosed with Parkinson's Disease by a neurologist
* Continuing anti-parkinsonian medication
* Hoehn-Yahr (H-Y) stage 3 and below
* Ability to walk independently
* To have full range of motion in shoulder abduction and elbow extension movements

Exclusion Criteria:

* Presence of additional neurological diseases other than Parkinson's Disease
* Scores below 21 on the Montreal Cognitive Assessment Scale
* Change in medication dosage in the last 1 month
* Severe visual impairment or complete hearing impairment in both ears
* Having a rheumatologic, musculoskeletal, etc. disease that may affect upper extremity functions
* The occurrence of severe tremors or dyskinesias due to the end of the drug dose
* Failing the Titmus butterfly test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test | through study completion, an average of 1 year
  The 19-item performance test will be used to assess the upper extremity function of the patients. The test is divided into four subscales: gross grasp, fine grasp, fingertip grip and gross movement. It is organized hierarchically from the most difficult task to the least difficult task. Task performance is assessed on a 4-point scale ranging from 0 (no movement) to 3 (movement is performed normally). Each section starts with the activity with the highest level of difficulty. If the individual can perform this activity without any problems, he/she gets full points from the other items in the section and moves on to the next section. The score ranges from 0-57 and low scores indicate that upper limb function is affected.
Proprioception Assessment | through study completion, an average of 1 year
  Position, i.e. proprioceptive sensation, will be evaluated with the "angle repetition test", one of the methods commonly used in the clinic. The person will be positioned in a sitting position with his/her back unsupported and feet touching the floor. The angle repetition test will be performed with a mobile device fixed above the elbow and between the shoulder. The person's eyes will be closed during the assessment to prevent the learning effect and the use of visual reference. After the shoulder is brought to the reference angle, the person is allowed to perceive the angle by waiting 10 seconds. The person will then be asked to bring his/her shoulder to the side of his/her body and then repeat the taught reference angle as he/she perceived it. The absolute value of the angle deviated from the target will be recorded. Measurements in the shoulder joint will be made at 40° and 100° angles.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | through study completion, an average of 1 year
  It is the most frequently used, valid and reliable scale for the assessment of impairments and disabilities in PD. It contains 42 items, consists of 4 sections and assesses patients' mental status, behavior and mental state (4 items), activities of daily living (13 items), motor functions (14 items) and treatment complications (11 items), respectively. Mental status; 16 points, activities of daily living; 52 points, motor functions; 108 points and treatment complications; 23 points, totaling 199 points. Higher scores indicate worsening of the patient's condition. An 8-point change in the total score was found to determine minimal clinically significant change.
Disabilities of the Arm, Shoulder, and Hand Questionnaire | through study completion, an average of 1 year
  It is a questionnaire consisting of a total of 30 questions used to evaluate the ability of the patient with upper extremity problems in activities of daily living and upper extremity functions. The first 21 questions ask about the degree of difficulty in performing various activities of daily living with the dominant limb in the last week, the next 5 questions ask about the degree of pain, numbness, weakness during activities and the last 4 questions ask about the effect of pathologies on sleep, work, social life and psychological status. For each question, the patient marked the appropriate response on a 5-point Likert-type scale. 1 indicates no difficulty, 2 indicates mild difficulty, 3 indicates moderate difficulty, 4 indicates extreme difficulty, and 5 indicates no difficulty at all. The questionnaire is evaluated between 30 and 150 points.
Parkinson's Disease Questionnaire (PDQ-8) | through study completion, an average of 1 year
  The questions in the PDQ-8 assess the condition of the individual in the last 1 month and are scored between 0 (never) and 4 (always). The total score is converted to a 100-point system and a high score indicates a decrease in quality of life.
Global rating of change score-GRC | average 1 year after the completion of the study
  It is a scale designed to determine the amount of improvement or deterioration of the patient over time. In our study, we will use the GRC version (-2: much worse, -1: worse, 0: same, 1: better, 2: much better), which consists of 5 levels between -2 and +2.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Kurul, Ph.D, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Faculty of Health Sciences Bolu Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No